CLINICAL TRIAL: NCT01600157
Title: Ambulant Laparoscopic Nephrectomy
Brief Title: Ambulant Laparoscopic Nephrectomy; Are There Limiting Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Nessn Azawi, senior urologist, Zealand University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SJ-267
Record Dates: First submitted 2012-05-12; First posted 2012-05-16 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Nephrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laparoscopic Nephrectomy (Experimental)
  Interventions: Procedure: Ambulant laparoscopic nephrectomy

INTERVENTIONS:
Procedure: Ambulant laparoscopic nephrectomy — The patients with a renal cancer diagnosis with be schedule to enter the project if they meet the inclusion criteria of the project and the postoperative period will be recorded to identified the limiting factors for ambulant laparoscopic nephrectomy.

SUMMARY:
Background Fast-track concepts reduced hospital stay from 15-20 days to three days for patients who underwent a colon resection [1-5]. A well-designed pilot study determined the efficacy of a fast-track program for a laparoscopic radical nephrectomy, and the fast-track group was discharged earlier from the recovery room median (74+/-23 v 103+/-47 minutes) as well as from the hospital median (41+/-11 v 59+/-11 hours) [6]. Implementation of the principles of the fast-track program shortened the postoperative hospital stay from eight to four days for patients who underwent an open radical nephrectomy [7]. Taek-Gu Lee et al. documented how early mobilization after colon surgery resulted in reduced recovery times without increased complications [8]. Laparoscopic surgery is minimal invasive with less surgical stress, morbidity and mortality [9]. The use of laparoscopic nephrectomy in Denmark reduces the hospital stay to 5.2 days which did not meet the foreign countries outcome [06].

Therefore a combination of the advantages of laparoscopic surgery and the fast-track concepts could be used by nephrectomies. However, no prospective studies describing the course after nephrectomies, where these advantages are exploited and it is important to make a basic study to describe and understand the factors of surgical outcome.

Aim of study To describe the postoperative period after laparoscopic trans-peritoneal nephrectomy that performed as an ambulatory procedure.

Method A prospective study will involve 62 patients who have been diagnosed with Cancer Renis DC649.

All patients will receive the results of CT-scanning at outpatient and of them who meet the inclusion criteria for the study will be informed about the study and will receive a written information according to appendix 1., and a new time with (NA) to get the results for kidney function and oral information about the study as well as their acceptation to be connected to the study, those patients will receive a standard recommendation to be discharged from hospital on the day of their operation and they will restart their normal activities the day after the operation unless there are preventing factors. All patients will be thoroughly informed by the examiner how to complete the questionnaire and will come through different tests according to appendix 2., a blood test will be taken according to appendix 12.

All patients should have a CT-scanning of abdomen, chest X-ray and kidney function test before the operations.

Statistic The number of patients, have been decided to be included to each study, is based on the realized number of nephrectomy operations that can be done during the specified period within each department and not on the statistic power of study.

The Scheffé's test will be used for multiple comparisons. The correlation between variables will be evaluated by using the Spearman's rank correlation coefficient. P values less than 0.05 is considered significant. Statistical analyses will be performed by SPSS statistic program software.

Publications The results of each study, irrespective of whether these are positive or negative, will be published in international scientific journals and will be distributed at relative conferences. The published articles will have Azawi NH as first author, Christensen T as last author and co-authors according to Vancouver rules.

Ethics The study will be reported to the Danish National Committee on Biomedical Research Ethics and regionsjaelland paraplygodtkendelsen data control, Ph.D. student (NA) will apply for enrollment to the PhD programme at the University of Copenhagen. Consent forms will be received from all patients and they will receive written information about project. The project will protect all of the data gathered.

ELIGIBILITY:
Inclusion Criteria:

1. Patient between 30-70 years old.
2. Diagnosed as Cancer Renis
3. Can read and understand Danish
4. No cardiac disease
5. No metastatic disease

Exclusion Criteria:

1. Mentally sick patient
2. Dement
3. Living alone
4. Cardiac problem
5. Multiple surgery previously
6. Per operative bleeding with the need to blood transfusion
7. Operation time at afternoon

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Identification of the limiting factors for ambulant laparoscopic nephrectomy | 8 hours
  The patient will asked a direct question after the operation if they can not be discharged at the operation day. what is the main reason not to be discharged at this time?
Identification of the limiting factors for ambulant laparoscopic nephrectomy | 1 day
  The patient will asked a direct question after the operation if they can not be discharged at the operation day. what is the main reason not to be discharged at this time?
Identification of the limiting factors for ambulant laparoscopic nephrectomy | 2 day
  The patient will asked a direct question after the operation if they can not be discharged at the operation day. what is the main reason not to be discharged at this time?
Identification of the limiting factors for ambulant laparoscopic nephrectomy | 3 day
  The patient will asked a direct question after the operation if they can not be discharged at the operation day. what is the main reason not to be discharged at this time?
Identification of the limiting factors for ambulant laparoscopic nephrectomy | 4 day
  The patient will asked a direct question after the operation if they can not be discharged at the operation day. what is the main reason not to be discharged at this time?

SECONDARY OUTCOMES:
Pain,Nausea,Vomiting,Fatigue,Dizziness | 3 hours
  The postoperative period of 30 days will be observed by using visual analog skala (VAS)for Pain,Nausea,Vomiting,Fatigue,Dizziness.
Pain,Nausea,Vomiting,Fatigue,Dizziness | 8 hours
  The postoperative period of 30 days will be observed by using visual analog skala (VAS)for Pain,Nausea,Vomiting,Fatigue,Dizziness.
Pain,Nausea,Vomiting,Fatigue,Dizziness | 1 day
  The postoperative period of 30 days will be observed by using visual analog skala (VAS)for Pain,Nausea,Vomiting,Fatigue,Dizziness.
Pain,Nausea,Vomiting,Fatigue,Dizziness | 2 day
  The postoperative period of 30 days will be observed by using visual analog skala (VAS)for Pain,Nausea,Vomiting,Fatigue,Dizziness.
Pain,Nausea,Vomiting,Fatigue,Dizziness | 3 day
  The postoperative period of 30 days will be observed by using visual analog skala (VAS)for Pain,Nausea,Vomiting,Fatigue,Dizziness.
Pain,Nausea,Vomiting,Fatigue,Dizziness | 4 day
  The postoperative period of 30 days will be observed by using visual analog skala (VAS)for Pain,Nausea,Vomiting,Fatigue,Dizziness.
Pain,Nausea,Vomiting,Fatigue,Dizziness | 5 day
  The postoperative period of 30 days will be observed by using visual analog skala (VAS)for Pain,Nausea,Vomiting,Fatigue,Dizziness.
Pain,Nausea,Vomiting,Fatigue,Dizziness | 10 day
  The postoperative period of 30 days will be observed by using visual analog skala (VAS)for Pain,Nausea,Vomiting,Fatigue,Dizziness.
Pain,Nausea,Vomiting,Fatigue,Dizziness | 30 day
  The postoperative period of 30 days will be observed by using visual analog skala (VAS)for Pain,Nausea,Vomiting,Fatigue,Dizziness.

CONTACTS AND LOCATIONS:
Overall Officials: Nessn Htum Azawi, M.D., Principal Investigator — Zealand University Hospital
Locations (1):
- Roskilde Hospital, Roskilde, Denmark

REFERENCES:
- [Background] Larson DW, Batdorf NJ, Touzios JG, Cima RR, Chua HK, Pemberton JH, Dozois EJ. A fast-track recovery protocol improves outcomes in elective laparoscopic colectomy for diverticulitis. J Am Coll Surg. 2010 Oct;211(4):485-9. doi: 10.1016/j.jamcollsurg.2010.05.007. Epub 2010 Aug 8. PMID 20822739
- [Background] Basse L, Jacobsen DH, Billesbolle P, Kehlet H. Colostomy closure after Hartmann's procedure with fast-track rehabilitation. Dis Colon Rectum. 2002 Dec;45(12):1661-4. doi: 10.1007/s10350-004-7255-0. PMID 12473891
- [Background] Basse L, Thorbol JE, Lossl K, Kehlet H. Colonic surgery with accelerated rehabilitation or conventional care. Dis Colon Rectum. 2004 Mar;47(3):271-7; discussion 277-8. doi: 10.1007/s10350-003-0055-0. PMID 14991487
- [Background] Hjort Jakobsen D, Sonne E, Basse L, Bisgaard T, Kehlet H. Convalescence after colonic resection with fast-track versus conventional care. Scand J Surg. 2004;93(1):24-8. doi: 10.1177/145749690409300105. PMID 15116815
- [Background] Nygren J, Hausel J, Kehlet H, Revhaug A, Lassen K, Dejong C, Andersen J, von Meyenfeldt M, Ljungqvist O, Fearon KC. A comparison in five European Centres of case mix, clinical management and outcomes following either conventional or fast-track perioperative care in colorectal surgery. Clin Nutr. 2005 Jun;24(3):455-61. doi: 10.1016/j.clnu.2005.02.003. Epub 2005 Apr 9. PMID 15896433
- [Background] Recart A, Duchene D, White PF, Thomas T, Johnson DB, Cadeddu JA. Efficacy and safety of fast-track recovery strategy for patients undergoing laparoscopic nephrectomy. J Endourol. 2005 Dec;19(10):1165-9. doi: 10.1089/end.2005.19.1165. PMID 16359206
- [Background] Firoozfard B, Christensen T, Kristensen JK, Mogensen S, Kehlet H. Fast-track open transperitoneal nephrectomy. Scand J Urol Nephrol. 2003;37(4):305-8. doi: 10.1080/00365590310014742. PMID 12944188
- [Background] Lee TG, Kang SB, Kim DW, Hong S, Heo SC, Park KJ. Comparison of early mobilization and diet rehabilitation program with conventional care after laparoscopic colon surgery: a prospective randomized controlled trial. Dis Colon Rectum. 2011 Jan;54(1):21-8. doi: 10.1007/DCR.0b013e3181fcdb3e. PMID 21160309
- [Background] Nishiguchi K, Okuda J, Toyoda M, Tanaka K, Tanigawa N. Comparative evaluation of surgical stress of laparoscopic and open surgeries for colorectal carcinoma. Dis Colon Rectum. 2001 Feb;44(2):223-30. doi: 10.1007/BF02234297. PMID 11227939